CLINICAL TRIAL: NCT07013916
Title: Fructose is a Metabolic and Inflammatory Pathogenic Factor in Metabolic Dysfunction-associated Steatohepatitis (MASH)
Acronym: FLOURISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: King's College London (Other); University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 344872
Record Dates: First submitted 2025-04-28; First posted 2025-06-10 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: MASH - Metabolic Dysfunction-Associated Steatohepatitis; MASH With Fibrosis; Steatosis of Liver
Keywords: fructose; MASH; MASLD; liver; inflammation
MeSH Terms: conditions — Fatty Liver; Inflammation | interventions — Fructose; Glucose

STUDY DESIGN:
Intervention Model Description: This is a four-week randomised double-blind parallel-arm food supplement intervention study that will determine the effect of fructose (arm 1) and glucose (arm 2) on metabolism in people with MASH (n=36), compared to people with simple steatosis (n=18), or controls without liver disease (n=18).
Who Masked: Participant, Investigator
Masking Description: Both participants and members of the research team will be blinded to the intervention allocation (fructose or glucose). The randomisation list will be maintained by an independent researcher with no role in conducting the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fructose supplementation (Active Comparator): Participants will consume 100 g/day of fructose powder administered as two 50g sachets, dissolved in water in addition to following a low-sugar diet
  Interventions: Dietary Supplement: fructose
- Glucose supplementation (Active Comparator): Participants will consume 100 g/day of glucose powder administered as two 50g sachets, dissolved in water in addition to following a low-sugar diet
  Interventions: Dietary Supplement: glucose

INTERVENTIONS:
Dietary Supplement: fructose — Fructose powder
  Arms: Fructose supplementation
Dietary Supplement: glucose — Glucose powder
  Arms: Glucose supplementation

SUMMARY:
MASLD (Metabolic dysfunction-associated steatotic liver disease) is a condition where fat builds up in the liver. It is the most common cause of liver disease worldwide. In some people, the fat can irritate the liver (inflammation) and cause damage. This is a more serious condition called MASH (Metabolic dysfunction-associated steatohepatitis). People with MASH more at risk of liver cirrhosis (advanced scarring in the liver) and liver cancer.

It is not fully understood why MASLD becomes MASH, or why this happens in some people but not in others. However, it is known that our diet plays a role. Research shows a diet high in a type of sugar called fructose might make MASLD worse. Fructose is found in fruit, honey and table sugar, and lots of processed food and drinks. The body deals with fructose differently to other sugars, which is why fructose may be a problem. Although scientists have studied the effects of fructose in healthy people, no studies so far have included people with MASH, so it is not known if fructose might make the condition worse.

To answer this question, the researchers will conduct a four-week randomised, double-blind study to compare the effects of fructose with another sugar called glucose in 36 people with MASH, 18 people with 'simple' MASLD, and 18 controls without liver disease. Participants will follow a low-sugar diet and, after 14 days on this diet, they will add either a glucose or fructose supplement for another 14 days. Participants will attend 3 study visits, where blood, urine, stool, and saliva samples will be taken. The main question is whether fructose causes more inflammation in people with MASH compared to those with MASLD, or people without liver disease. The researchers will also investigate how fructose affects liver fat content, the gut microbiota, and other processes relevant to MASLD/MASH.

DETAILED DESCRIPTION:
Overview of the study:

This is a four-week randomised double-blind parallel-arm food supplement intervention study that will determine the effect of fructose on metabolism in people with MASH, compared to people with simple steatosis, or controls without liver disease. The study will involve consent (visit 0A) and screening (visit 0B), followed by two study stages (see Figure 1), where participants will undergo study visits and procedures as detailed in Table 1. Each participant will attend for a total of up to 5 study visits: consent (visit 0A) and screening (visit 0B); Baseline (visit 1); pre-intervention (visit 2); post-intervention (visit 3). Consent (visit 0A) and screening (visit 0B) visits may be combined into one visit if feasible and the participant would like to do so. Otherwise, visits will be conducted on separate days as close together as practical for the participant and research team (ideally no more than 3-4 weeks). Visits 1 to 3 will each last approximately 8 hours, at which participants will consume a test meal and have hourly blood samples taken via a cannula for approximately 6h.

A subset of participants (maximum of n=24; n=12 MASH; n=12 steatosis/control) will be invited to take part in an optional sub-study. This will involve the same study visits and procedures as the main study but will additionally measure how glucose or fructose is metabolised in the postprandial state by addition of a small amount of glucose/fructose stable isotope tracer (13C6-fructose or 13C6-glucose) to the metabolic test meal. Participants will also provide breath samples at hourly intervals during the 6h feeding period.

There will be no change to routine patient care for MASH and MASLD participants during the study period. Any clinically significant results emerging from study participation will be shared with participants' GP or care team.

Description of the study intervention:

Following consent (visit 0A) and screening (visit 0B), participants will receive a study guide with details of the main study visits and procedures, and instructions on how to complete the 3-day food diaries. At the baseline visit (visit 1), participants will receive dietary counselling and other information to help them follow a diet low in free sugars, including fructose, glucose, and sucrose. The nutrition researcher and participant will agree on a personalised list of suggested low-sugar meals, drinks and snacks that are suitable to be consumed during the study. Participants will be given a choice of food, drink and snack items to be delivered each two weeks as the basis for a low-sugar diet. The nutrition researcher will offer ongoing support to ensure compliance via regular phone calls, messages, and at study visits as needed.

Following the Baseline visit (visit 1), participants will undergo a two-week run-in period on the low-sugar diet, after which they will be randomised to either group A or B for the supplementation period. Both groups will be maintained on the low-sugar diet and additionally receive supplemental 100g of fructose (group A) or glucose (group B) per day for a period of 14 days. All sachets will be labelled as 'Sugar Supplement' or similar.

Each 100g daily dose of glucose or fructose will be prepared by an independent researcher at King's College London and divided into two labelled sachets (50g each). Participants will be directed to dissolve each of the sugar sachets in approximately 300 ml of water and to consume these solutions in between their primary meals. All study participants will be provided with a daily multivitamin supplement to prevent any risk of nutrient deficiencies due to the low fruit content of the prescribed diet.

Dietary intake will be analysed through a series of 3-day food diaries completed contemporaneously prior to each of the study visits (baseline, pre- and post-intervention). The UK Composition of Foods Integrated Dataset will be used to compute the macro- and micronutrient composition, as well as the caloric value, of the diet. The dietary intervention will be compiled by an expert nutrition researcher and overseen by a qualified dietitian.

Participants will attend five study visits, including consent (visit 0A) and screening (visit 0B), a baseline visit (visit 1; before starting the low-sugar diet), as well as visits pre-intervention (visit 2) and post-intervention (visit 3), as detailed in section 7.3. Consent (visit 0A) and screening (visit 0B) visits may be combined into one visit if feasible and the participant would like to do so.

Participants will be remunerated for their time and commitment to completing the study procedures.

Visits for the study:

Pre-screening: Potential participants will be recruited from liver clinics (MASH and steatotic patients) or via the PIC site (King's College Hospital); control (healthy) participants will be recruited via email or poster adverts. All potential participants will receive a copy of the Participant Information Sheet and be given time to read and consider this. Prior to attending for a consent or screening visit, potential participants will undergo a pre-screening call or discussion with either a member of their clinical care team (MASH/steatosis patients) or a member of the study research team (controls) to check their eligibility against the inclusion/exclusion criteria prior to attending in person.

Consent (Visit 0A): Prior to the consent visit, participants will receive the participant information sheet and have the opportunity to consider this (and discuss it with others if they wish). Participants will attend for the visit and have the opportunity to ask questions or discuss the study with a member of the research team, before offering their informed consent. Participants will receive a copy of their signed consent form and agree on a suitable date for the screening visit.

Screening (visit 0B): Participants will answer questions concerning medical history, have anthropometrics and vital signs measured by a researcher, and (if required to confirm eligibility) have a Fibroscan and fasted blood sample taken. Participants will be informed of their eligibility following the visit and be provided with a copy of the study guide, which includes instructions on how to complete the 3-day food diaries.

Visits 1, 2 and 3: Participants will be sent a reminder to complete each of the 3-day food diaries prior to each visit. They will also be given a low-fat standardised meal to consume the night before and will attend in the morning (at approximately 8am) after an overnight fast (≥12h). Participants will provide fresh stool, urine, and saliva samples, and researchers will take anthropometric measurements and vital signs (e.g. blood pressure). Measurements will be conducted utilising Vibration-Controlled Transient Elastography with Controlled Attenuation Parameter (VCTE CAP).

Participants will then undergo a 6-hour post-prandial feeding protocol, which will measure the metabolic response to consuming a standardised mixed nutrient test meal. Participants will be cannulated and have fasted blood samples taken, before consuming the mixed-nutrient meal. Blood samples will be taken every hour over the subsequent 6-hour period to test metabolic response to the test meal, including markers of lipid and glucose metabolism. Participants will not be able to eat anything else during this period but will be offered ad libitum drinking water.

In the optional sub-study, participants will additionally consume 13C6-glucose or 13C6-fructose stable isotope tracer as part of the test meal and provide breath samples at hourly intervals, in addition to the hourly blood samples. This will allow the metabolism of glucose and fructose to be measured in blood (13C-palmitate for de novo lipogenesis) and breath (13CO2 for glucose/fructose oxidation) samples to provide additional insight into how the sugars are metabolised.

Following the post-prandial procedure, the cannula will be removed. Participants will be offered something to eat, given any additional instructions, dietary counselling, or study supplies required for the next stage of the study and will then be able to leave.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent
* Age 45-65 at consent
* HbA1c < 48 mmol/mol
* Overweight and stage I obesity using BMI thresholds adjusted for ethnicity:

  * 23.0kg/m2 - 32.4kg/m2 in South Asian, Chinese, other Asian, Middle Eastern, Black African or African-Caribbean populations
  * 25kg/m2 - 34.9kg/m2 in White populations

MASH Patients:

Clinical diagnosis of MASH and F2 - F3 fibrosis:

Either:

Liver biopsy within 12 months of baseline

Or:

• History of histologically-diagnosed MASH with current evidence of fatty liver, AST>20 and Fibroscan CAP≥248 dB/m and stiffness 9.5kPa -14kPa

Or:

• FAST score >0.67

Patients with steatosis:

• defined by Fibroscan CAP≥248dB/m and stiffness <7.9kPa.

Healthy controls:

• defined by Fibroscan CAP<248dB/m and stiffness <7.9kPa.

Exclusion Criteria:

* Unwilling or unable to give consent
* Age <45 or >65
* Any form of diabetes mellitus
* Currently pregnant
* Known fructose intolerance or food allergy
* Diagnosis of cirrhosis or Fibroscan stiffness >14kPa
* Current Child-Pugh B/C or episode of decompensation in last year
* Non-MASLD liver disease known to participant (including viral hepatitis, auto-immune hepatitis, primary sclerosing cholangitis, primary biliary cholangitis, haemochromatosis, sarcoidosis, cystic fibrosis, sickle cell disease)
* Regular alcohol intake > 14 units a week for females and >21 units a week for males (participant-reported)
* Smoking, vaping or use of nicotine-containing products within the last month
* Taking prohibited medication:

  * Probiotic or antibiotic use within last 4 weeks (Note: participants will be considered eligible if they have undergone a 4-week washout from probiotics or 4-weeks after discontinuing antibiotic use)
  * any oral steroids within the last 6 weeks
  * current, or within 3 months, use of immunosuppressive medication
  * Amiodarone, nitrofurantoin, or anti-fungals within 3 months
  * Use of anti-obesity medication - orlistat or GLP-1 receptor agonist-containing treatments within 6 months
  * Use of vitamin E, pioglitazone or other medication for MASH including current or within 3 months enrolment in clinical trial unless documented to have been on placebo
* History of malignancy (except basal cell carcinoma), or medication for malignancy within the last 2 years
* Any major organ transplant (excluding corneal or hair)
* Clinical diagnosis of chronic kidney disease 3 or above, or of heart failure (NYHA 3 or 4)
* COPD requiring home oxygen
* Known eating disorder (e.g. anorexia nervosa) or severe mental illness (e.g. schizophrenia)
* Investigator opinion that study is unsuitable for patient

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in plasma glutamate concentration | Changes from baseline to week 2
  Difference in the fructose-induced changes in plasma glutamate concentration in patients with MASH and fibrosis compared to patients with simple steatosis (without fibrosis) or healthy controls.

SECONDARY OUTCOMES:
Plasma metabolome | Changes from baseline to week 2
  Changes in plasma metabolome from blood samples measured by mass spectrometry
Urine metabolome | Changes from baseline to week 2
  Changes in urine metabolome measured by mass spectrometry
Plasma glucose | Changes from baseline to week 2
  Changes in fasting and post-prandial plasma glucose (mmol/L)
Plasma triglycerides | Changes from baseline to week 2
  Change in fasting and post-prandial plasma triglycerides (mmol/L)
Serum insulin | Changes from baseline to week 2
  Change in fasting and post-prandial serum insulin (pmol/L)
De novo lipogenesis | Changes from baseline to week 2
  Change in absolute fasting and post-prandial de novo lipogenesis measured as 13C-palmitate in plasma triglyceride-rich lipoproteins (µmol/L)
Liver function markers | Changes from baseline to week 2
  Changes in liver function enzymes (ALT, AST, ALP, GGT), albumin and bilirubin
Gut hormones | Changes from baseline to week 2
  Changes in hormones relevant to gut function (e.g. digestion) and/or physiology, measured using standardised tests.
Oral microbiome | Changes from baseline to week 2
  Changes in oral microbiome measured from saliva samples using 16S sequencing
Oral metabolites | Changes from baseline to week 2
  Changes in metabolites from saliva samples measured using mass spectrometry
Markers of inflammation | Changes from baseline to week 2
  Changes in markers of inflammation
Markers of immunity | Changes from baseline to week 2
  Changes in markers of immune function
Markers of cell function | Changes from baseline to week 2
  Changes in markers of cell function

OTHER OUTCOMES:
Genetic variants | Changes from baseline to week 2
  Measures of genetic variants relevant to MASLD/MASH and/or relevant metabolic processes, including sugar digestion/metabolism, inflammation, and/or liver metabolism.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal London Hospital, London
  - Blizard Institute, Faculty of Medicine and Dentistry, Queen Mary University of London, London

IPD SHARING:
Plan to Share IPD: No